CLINICAL TRIAL: NCT06920420
Title: Xuebijing Injection Regulates Endothelial Cell Panapoptosis in Treating Sepsis Through PCDHAC2/BAX/AIM2 Pathway
Brief Title: Novel Biomarkers Related Xuebijing Injection Improves Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Prof, Southeast University, China
Other Study IDs: 2024ZDSYLL513-P01; 82472202 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Xuebijing treatment group: Based on the standard treatment group Xuebijing injection was added.
- Standard treatment group: Patients with sepsis are given standard treatment according to international guidelines for the management of sepsis and septic shock
- Healthy Volunteer Group

SUMMARY:
Sepsis is a life-threatening clinical syndrome of organ dysfunction caused by dysregulation of the body's response to infection, and is a common cause of ICU admission for critically ill patients, posing a serious threat to human health. The study demonstrated that hemopexin injection significantly reduced the 28-day all-cause mortality rate of sepsis patients, and this study clarified the specific target and molecular mechanism of hemopexin injection in the treatment of sepsis, which may be of great scientific significance and clinical value for the precise treatment of sepsis and the research and development of new drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the Sepsis 3.0 diagnostic criteria;
2. SOFA score ≥ 2 and < 13;
3. Signed informed consent.

Exclusion Criteria:

1. Age <18 years or >75 years;
2. Pregnant or lactating women;
3. Presence of severe primary diseases including malignant tumors severe hematologic disorders and HIV infection;
4. Current use of immunosuppressants or history of organ transplantation within the past 6 months;
5. Comorbidities that significantly affect vascular endothelial structure and function such as acute myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sepsis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Single-cell transcriptomic analysis of inflammatory and metabolic gene expression, measured using scRNA-seq, with data summarized as differential expression profiles. | Day7
  Single-cell transcriptomic analysis of inflammatory and metabolic gene expression, measured using scRNA-seq, with data summarized as differential expression profiles.

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data, including genetic information, will not be shared due to privacy and ethical considerations. Genetic data is highly sensitive and could potentially identify individuals. To protect patient confidentiality and comply with regulations such as GDPR and HIPAA, access to such data is strictly limited and will only be shared under explicit informed consent and approved ethical guidelines.